CLINICAL TRIAL: NCT02077322
Title: Rates of Middle Meatal Synechia Formation Following Functional Endoscopic Sinus Surgery: A Double-Blind Randomized Controlled Trial Comparing Gloved Merocel and Silastic Middle Meatal Spacers.
Brief Title: Rates of Middle Meatal Synechia Formation Following Functional Endoscopic Sinus Surgery
Acronym: SYNECHIAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Synechiae-2014
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Sinusitis
Keywords: Merocel Middle Meatus Spacers; Silastic Middle Meatus Spacers; Functional Endoscopic Sinus Surgery
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silastic Spacer (Experimental): This study arm receives the experimental treatment, a Silastic spacer.
  Interventions: Device: Silastic Spacer
- Merocel Spacer (Active Comparator): Merocel spacers are actively being used as the standard of care.
  Interventions: Device: Merocel Spacer

INTERVENTIONS:
Device: Silastic Spacer — The Silastic spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6 to 14 days following surgery.
  Other Names: Experimental Arm
  Arms: Silastic Spacer
Device: Merocel Spacer — The Merocel spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6 to 14 days following surgery.
  Other Names: Control Arm
  Arms: Merocel Spacer

SUMMARY:
Functional endoscopic sinus surgery (FESS) is the best method of surgically treating patients who suffer from sinus disease. Synechiae formation in the nose is the most common complication after sinus surgery. Synechiae describes the adhesion of two opposing mucosal surfaces in the nasal cavity that can cause scarring and obstruction of the nasal passage. Spacers are often inserted during surgery between nasal mucosal surfaces to prevent synechiae. The aim of this study is to see if a silastic spacer is more effective at reducing the formation of synechiae after sinus surgery than a merocel spacer.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 19 years, currently receiving sinus-related care at the St Paul's Sinus Centre for chronic rhinosinusitis and who undergo primary bilateral complete endoscopic sinus surgery will be approached to participate in this clinical trial.

Exclusion Criteria:

* Patients with sino-nasal tumors
* Patients solely undergoing nasal septal reconstruction
* Patients with previous history of endoscopic sinus surgery
* Cystic fibrosis or syndromic patients
* Patients with autoimmune diseases

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Incidence of middle meatal synechiae after functional endoscopic sinus surgery in silastic versus merocel groups. | Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
  The existence of postoperative synechiae will be considered as a categorical, dichotomous outcome variable (presence or absence). A senior Rhinologist will endoscopically assess each nasal cavity independently to determine if synechiae exists between the middle turbinate and lateral nasal wall. Count and absolute percentages will be reported.
  Incidence of postoperative synechiae will be compared between right and left nasal cavities receiving either silastic or glove finger spacers.

SECONDARY OUTCOMES:
Incidence of postoperative synechiae in 6-day versus 14-day postoperative spacer removal groups. | Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
  The existence of postoperative synechiae will be considered as a categorical, dichotomous outcome variable (presence or absence). A senior Rhinologist will endoscopically assess each nasal cavity independently to determine if synechiae exists between the middle turbinate and lateral nasal wall. Count and absolute percentages will be reported.
  Secondary comparisons of postoperative synechiae will be compared between subjects in the 6-day vs 14-day spacer removal groups.

OTHER OUTCOMES:
Sinonasal Outcomes Test-22 (SNOT- 22) score. | Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
  The SNOT-22 is a sinus-specific questionnaire that evaluates subjective symptoms for patients suffering from chronic rhinosinusitis. SNOT-22 is scored out of 110 (22 questions, up to 5-points each) has demonstrated internal consistency, reliability, discriminate and concurrent validity and responsiveness to change12. Responses will be summated and considered as a continuous, numerical variable. Mean, median, standard deviation and inter-quartile range will be reported.
  SNOT-22 change between baseline (preoperative score) and 90-days (postoperative score) will be compared between groups having middle meatal spacers removed at 14 days versus 6 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD, FRCSC, FARS, Principal Investigator — St. Paul's Hospital, Canada
Locations (1):
- St. Paul's Hospital Sinus Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Miller RS, Steward DL, Tami TA, Sillars MJ, Seiden AM, Shete M, Paskowski C, Welge J. The clinical effects of hyaluronic acid ester nasal dressing (Merogel) on intranasal wound healing after functional endoscopic sinus surgery. Otolaryngol Head Neck Surg. 2003 Jun;128(6):862-9. doi: 10.1016/S0194-59980300460-1. PMID 12825038
- [Background] Catalano PJ, Roffman EJ. Evaluation of middle meatal stenting after minimally invasive sinus techniques (MIST). Otolaryngol Head Neck Surg. 2003 Jun;128(6):875-81. doi: 10.1016/S0194-59980300469-8. PMID 12825040
- [Background] Lee JM, Grewal A. Middle meatal spacers for the prevention of synechiae following endoscopic sinus surgery: a systematic review and meta-analysis of randomized controlled trials. Int Forum Allergy Rhinol. 2012 Nov;2(6):477-86. doi: 10.1002/alr.21052. Epub 2012 May 30. PMID 22648984